CLINICAL TRIAL: NCT02550626
Title: Exploring the Relationship Between Alpha-synucleinopathy Related Non-motor Symptom and Post-op. Delirium in Elderly Patients With Spine Surgery
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-0365
Record Dates: First submitted 2015-07-16; First posted 2015-09-15 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Post-operation Delirium; Alpha-synucleinopathy Related Non-motor Symptom
Keywords: delirium; alpha synucleinopathy; spine surgery
MeSH Terms: conditions — Delirium; Synucleinopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Delirium: occurrence of post-operative delirium
- No delirium: no presence of post-operative delirium

SUMMARY:
Hypothesis is that the presence of a-synucleinopathy related non motor symptoms could be predictive factor for post-operative delirium. During 72hrs after spine surgery, investigator will observe occurrence of post-operative delirium, and analysis difference of a-synucleinopathy related non motor symptoms between 2 groups.

DETAILED DESCRIPTION:
Postoperative delirium appear approximately 10-70% of patients older than 65 yrs undergoing surgery and it is strongly associated with poor surgical outcome. The clinical characteristics of postoperative delirium are fluctuating attention, visual hallucination, disorganized thought and alter sleep-wake cycles. This is quite similar to core features of α-synuclein-related cognitive disorders such as parkinson's disease dementia and dementia with lewy body. At that point, investigator thought that postoperative delirium is preclinical stage of a-synucleinopathy. In other words, a-synuclein related disorders and postoperative delirium may share an underlying neurochemical change in their pathogenesis.

investigator will recruit age 65 and older patients scheduled to perform spine surgery. The pre-operative evaluation include neurologic exam, baseline cognitive function and a-synucleinopathy related non motor symptoms through Questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 and older patients
2. Scheduled to perform spine surgery in severance hospital

Exclusion Criteria:

1. Previous delirium history
2. Previous chemotherapy or radiotherapy within 1yr due to underlying cancer.
3. Severe hepatic/renal dysfunction

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: spine surgery
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
existence of anosomia | A day before operation
  During 72hrs after spine surgery, investigator will observe occurrence of post-operative delirium, and analysis difference of anosmia symptoms before operation between 2 groups. The cross-cultural smell identification test will be used for measure of anosmia. investigator define anosmia as less than 4 score on the cross-cultural smell identification test. This study is not interventional study, because measure of anosmia by smell kit will not develop post-operation delirium more. (investigator will classify our patients into normosmia if the CCSIT score is 9 or higher, and hyposmia if the CCSIT score is 6 or less. Patients whose CCSIT scores are 7 or 8 will be regarded as borderline.).

SECONDARY OUTCOMES:
existence of constipation | A day before operation
  Questionnaire (Constipation scoring system (Agachanet al., 1996) & Rome III Questionnaire (Constipation : Yes/No)
existence of orthostatic hypotension | A day before operation
  Check 3 position BP (define orthostatic hypotension - sustained reduction of systolic blood pressure of at least 20 mmHg or diastolic blood pressure of 10 mmHg within 3 min of standing, / Questionnaire (orthostatic hypotension symptom assessment & Orthostatic hypotension daily activities scale) (orthostatic hypotension: Yes/No)
existence of insomnia | A day before operation
  Questionnaire (Epworth Sleepiness Scale (ESS) : total score 0-24)
existence of depression | A day before operation
  Questionnaire (Beck depression inventory, total score 0-63)
existence of anxiety | A day before operation
  Questionnaire (The Parkinson Anxiety Scale, total score 0-48)
existence of REM sleep behavior disorder | A day before operation
  Questionnaire (RBD screening questionnaire, total score 0-13) :These questionnaires & checking 3-position BP will not effect the occurence of post-operation delirium

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Yonsei University College of Medicine, Seoul, Seou, South Korea